CLINICAL TRIAL: NCT02332694
Title: Whole Body Hyperthermia (WBH) as a Rapid Treatment for Fibromyalgia
Acronym: Fibro and WBH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator transferred to the University of Wisconsin - Madison
Sponsor: Charles (Chuck) Raison (Other)
Responsible Party: Sponsor-Investigator, Charles (Chuck) Raison, Professor, Department of Psychiatry; College of Medicine, University of Arizona
Organization: University of Arizona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #14-1261-1804
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High intensity whole-body infrared heating (Experimental): The participant will undergo the WBH intervention where subjects will be induced to levels of heat that increases core body temperature to approximately 37.5-38.5 °C.temperature.
  Interventions: Device: The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation

INTERVENTIONS:
Device: The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation — The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation. The rise in the body's core temperature is correspondingly rapid and well-tolerated. There are two phases of the thermal challenge, 1) Irradiation phase during which the patient lies recumbent with his/her head positioned outside the tent. The wIRA irradiators are arranged above the exposed upper part of the body; and 2) Heat retention phase during which the patient lies in the chamber with the walls of the tent positioned to retain heat. Core body temperatures will be raised to those comparable to a mild fever 37.8-38.5°C.

SUMMARY:
Fibromyalgia has become an increasingly pressing public health problem in the United States. Although some treatments exist for Fibromyalgia, many individuals suffering with Fibromyalgia do not adequately respond to currently available treatment options, highlighting the need to develop and test new interventions for the disorder. To address this pressing clinical issue, we will conduct a pilot study to determine if Whole Body Hyperthermia (WBH) reduces symptoms in adults suffering from Fibromyalgia. We plan to recruit individuals with Fibromyalgia who will receive a single session of WBH to determine if this single session improves Fibromyalgia symptoms and if so whether this improvement will last at least 2 weeks. To do this, the study will include self-report symptom assessments immediately before and one and two weeks after WBH. In addition blood will be collected at these time points to explore whether WBH changes immune system chemicals that are believed to contribute to fibromyalgia. We intend to conduct the study until 10 individuals with fibromyalgia have received a single treatment of WBH and have completed all pre-treatment and post-treatment assessments. Given scientific evidence from our research group that WBH may improve depression, we anticipate that it may also be of benefit or adults suffering from Fibromyalgia.

DETAILED DESCRIPTION:
We will direct a clinical trial of Whole Body Hyperthermia (WBH) for the treatment Fibromyalgia. Although we have not yet studied WBH for Fibromyalgia we have data indicating that WBH is effective for the acute treatment of major depression (MDD). Given the high overlap of symptoms between Fibromyalgia and Major Depressive Disorder (MDD), we have reasons for expecting that WBH may also be of benefit for Fibromyalgia. The primary objective of the proposed study is to determine if WBH produces improvement in core Fibromyalgia symptoms, just as it appears to do in MDD. Indeed, in preliminary studies, a single exposure to WBH resulted in a downward shift in body temperature (Figure 6) and a decrease in depressive symptoms as measured using the Center for Epidemiologic Studies Depression Scale (known as the ADS in Germany where this study was conducted) 5 days later (Figure 7). In addition, following exclusion of one patient with bronchopulmonary inflammation that did not show a decrease in body temperature following treatment, a correlation between the shift in body temperature and ΔADS approached statistical significance (Figure 9). These preliminary data are consistent with previous studies showing that 1) patients with seasonal affective disorder in winter during depression have blunted thermoregulatory cooling but have thermoregulatory cooling that is similar in efficiency to control subjects after successful antidepressant response to phototherapy (the retina has direct projections to DRVL serotonergic neurons), 2) ECT increases the circadian amplitude of core body temperature, and decreases mean core body temperature, particularly during the nighttime thermoregulatory cooling period, and 3) thermoregulatory cooling, as evidenced by the number of active sweat glands in depressed patients, increases upon clinical recovery, but not earlier, following ECT. We hypothesize that these relationships in preliminary data and in previous studies are due to dysfunction of the afferent signaling arm of the thermoregulatory system in MDD, specifically the warm afferent system projecting to the LPB and, secondarily, to the DRVL/VLPAG and DRI subsets of serotonergic neurons that have been implicated in anxiolytic and antidepressant actions, respectively, and to normalization of warm afferent signaling following treatment. Again given the high degree of overlap between Fibromyalgia and MDD, we expect that WBH may confer therapeutic benefits in Fibromyalgia as it appears to do in MDD.

This clinical trial will only include individuals with Fibromyalgia (i.e. no normal controls) in order to determine whether there is a significant effect of a single treatment with WBH administered in an open manner on Fibromyalgia symptoms. Based on our data from patients with MDD, we expect that if WBH has an effect on Fibromyalgia symptoms this will be apparent immediately after the treatment and will persist for at least a week. Therefore we will assess Fibromyalgia symptoms prior to and at 1 and 2 weeks following a single treatment with WBH. To evaluate whether treatment effects are longer lasting we will also assess symptoms two weeks following the WBH treatment.

Useful preliminary results were obtained from a pilot study comparing mildly to severely depressed patients receiving hyperthermic treatment (N=11) to depressed patients receiving psychotherapy as usual (N=3). Baseline scores on the German language ADS depression scale were similar for the two groups (mean=30.64, sd=9.18, N=11, vs. mean =32.33, sd=17.04, N=3). Raw change on the ADS was significantly greater for the hyperthermia group (mean=-11.91, sd=6.55, N=11, vs. mean=-1.33, sd=4.51, N=3; t=2.60, df=12, P=0.023), resulting in a very large standardized treatment difference (Cohen d) of 1.69 (95% CI=1.00 - 2.48). Percent change was also significant (mean=-39.4, sd=18.9, N=11, vs. mean=-8.6, sd=17.0, N=3; t=2.54; df=12, P=0.026), for a Cohen d of 1.66 (95% CI=0.93 - 2.39). The percentage of the hyperthermia vs. psychotherapy group achieving a clinical response (>50% reduction from baseline) was 27.3% vs. 0%, and the percentage achieving at least a partial response (>25% improvement) was 81.8% vs. 33.3%.

These data suggest that our proposed sample size of 10 individuals with Fibromyalgia should be sufficient to identify a potential therapeutic effect, assuming that such an effect would be of similar magnitude to the effect seen in MDD. To obtain a cohort of 10 subjects with complete baseline and post-treatment data we anticipate enrolling between 12 and 15 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* A diagnosis Fibromyalgia based on a clinician's diagnosis.
* In the investigator's opinion, has met criteria for Fibromyalgia for at least 4 weeks prior to signing consent.
* Able to communicate in English with study personnel.
* For women, must not be pregnant (per urine test)

Exclusion Criteria:

* Any of the following diagnoses, as identified by the psychiatric evaluation or study assessments:

  * A current DSM-IV-TR Axis I diagnosis of Dementia; or
  * Any current DSM-IV-TR Axis II diagnosis (i.e. personality disorder) that would suggest potential noncompliance with the protocol; or
  * A lifetime history of Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder Type 1; or
  * A diagnosis claustrophobia severe enough that it would impair ability to be in the Heckel HT3000 hyperthermia device
* A current (or within 12 months prior to the Screening visit) diagnosis of Anorexia Nervosa or Bulimia Nervosa
* Subject has met DSM-IV criteria for Substance Abuse in the month prior to screening visit
* A diagnosis of an anxiety or mood disorder that is considered by the investigator to be of greater source of distress or functional impairment than the patient's FIBROMYALGIA diagnosis. Subjects with comorbid anxiety and mood disorders not excluded above and considered to be of secondary importance will be permitted in the study.
* Participation in concurrent formal psychotherapy during the trial, or in the 2 weeks prior to the screening visit.
* Subject has a medical condition or disorder that:

  * Is unstable and clinically significant, or:
  * Could interfere with the accurate assessment of safety or efficacy of treatment, including:
  * individuals who are using prescription drugs that may impair thermoregulatory cooling, including diuretics, barbiturates, and beta-blockers, or antihistamines,
  * individuals with cardiovascular conditions or problems (uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease)
  * individuals with chronic conditions/diseases associated with a reduced ability initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy,
  * hemophiliacs/individuals prone to bleeding,
  * individuals with a fever the day of study intervention (if so, they will be rescheduled),
  * individuals with hypersensitivity to heat,
  * individuals with recent acute joint injury (i.e. arthritis),
  * individuals with enclosed infections, be they dental, in joints, or in any other tissues,
* Clinically significant, in the investigator's opinion, abnormal findings on screening laboratory tests or physical exam.
* Use of any psychotropic medications for 2 weeks (8 weeks for fluoxetine) prior to initiation of the study, with the exception of a stable dosage of benzodiazepine or non-benzodiazepine hypnotic medications (e.g. zolpidem (Ambien), zaleplon (Sonata), eszopiclone (Lunesta), lorazepam (Ativan), diazepam (Valium), clonazepam (Klonopin), alprazolam (Xanax),
* Need for any non-protocol psychotropic medication once enrolled, with the exception of benzodiazepine or non-benzodiazepine hypnotics used at a stable dosage.
* Women who are pregnant (HCG pregnancy test at screening, or lactating, or who plan to become pregnant during the study.
* Current participation in any clinical trial that might impact results of this one, which includes participation in another clinical trial, as well as drug trials with agents that might affect mood or regulation of body temperature or core fibromyalgia symptoms
* Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.
* Obesity and overall size of subject. It will be up to the PI's discretion to consider BMI, waist circumference, and body fat composition when determining eligibility and safety of the individual.
* History of peripheral circulatory disease, for example peripheral vascular disease, deep vein thrombosis (DVT), or lymphedema.
* History of a cerebral vascular accident
* History of stroke, epilepsy or cerebral aneurisms
* Cancer in the last five years, except for fully resected non-melanoma skin cancer.
* Diabetes mellitus types I or II.
* Any clinically significant autoimmune disease (compensated hypothyroidism allowed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The Fibromyalgia Impact Questionnaire (FIQ) | Screening, baseline and 1 and 2 weeks post-intervention
  Change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on fibromyalgia symptoms.

SECONDARY OUTCOMES:
The Brief Pain Inventory (BPI) | Screening, baseline and 1 and 2 weeks post-intervention
  Change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on fibromyalgia pain symptoms.
Change in depression scores over time [Inventory of Depressive Symptomatology-Self Report (IDS-SR)] | Screening, baseline and 1 and 2 weeks post-intervention
  Percent change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on depression symptoms.
Change in Scores on the Brief COPE Measure | Screening, baseline and 1 and 2 weeks post-intervention
  Percent change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on participant's ability to cope.
Change in Scores on the Sheehan Disability Scale (SDS) | Screening, baseline and 1 and 2 weeks post-intervention
  Percent change in scores between baseline and subsequent assessments will be assessed to assess functional impairments in three inter-related domains, work/school, social and family life.
Plasma Concentrations of Biological Predictors of Response and Mechanism of Action for WBH | Baseline and 1 and 2 weeks post-intervention
  Blood samples will be analyzed for physiological measures expected to be impacted by WBH including RNA expression, plasma concentrations of BDNF, and pro- and anti-inflammatory cytokines.
Change in Score on the Q-LESQ-SF (Quality of Life Enjoyment and Satisfaction Questionnaire -Short form) | Screening, baseline and 1 and 2 weeks post-intervention
  Percent change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on self-reported quality of life.
Change in Score on the Edinburgh Warwick Scale | Baseline and 1 and 2 weeks post-intervention
  Percent change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on positive emotions during the study
Change in Score on the Positive and Negative Association Scale (PANAS) | up to 2 weeks post-intervention
  Percent change in scores on the PANAS Scale to assess the transient and fluctuating active mood states during the WBH procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona, Department of Psychiatry, College of Medicine
Locations (1):
- University of Arizona, Tucson, Arizona, United States